CLINICAL TRIAL: NCT03866668
Title: An Open-Label Pilot Study of Esomeprazole in Children With Autism
Brief Title: A Study of Esomeprazole in Children With Autism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: SPARK (Stanford University) (Unknown)
Responsible Party: Principal Investigator, Antonio Hardan, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-44589
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Esomeprazole
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Esomeprazole (Experimental): Esomeprazole Dosage (Weight Less Than 20 kg) -- 10 mg QD for 8 weeks Esomeprazole Dosage (Weight 20 kg or Greater) -- 10 mg QD for 4 weeks followed by 20 mg QD for 4 weeks
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole Dosage (Weight Less Than 20 kg) -- 10 mg QD for 8 weeks Esomeprazole Dosage (Weight 20 kg or Greater) -- 10 mg QD for 4 weeks followed by 20 mg QD for 4 weeks
  Other Names: Nexium

SUMMARY:
Autism is a pervasive developmental disorder characterized by core deficits in social behavior and communication and the presence of repetitive/stereotyped behaviors. The objective of the study is to evaluate the efficacy of Esomeprazole as a treatment for social communication deficits in children with Autism Spectrum Disorder (ASD). This prospective 12 week open-label study will invite 25 children with ASD between the ages of 2 and 6 years of age to participate.

ELIGIBILITY:
Inclusion Criteria:

* outpatients 2 to 6 years of age;
* males and females who are physically healthy;
* diagnosis of autism spectrum disorder based on clinical evaluation and DSM-5 criteria, and confirmed using the Autism Diagnostic Interview-Revised, and the Autism Diagnostic Observation Schedule or Childhood Autism Rating Scale second edition (CARS-2)
* care provider who could reliably bring subject to clinic visits, could provide trustworthy ratings, and interacted with subject on a regular basis;
* ability of subject to swallow the compound;
* stable concomitant medications for at least 2 weeks (4 weeks if patient took fluoxetine);
* no planned changes in psychosocial interventions during the open-label trial.

Exclusion Criteria:

* DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder not otherwise specified;
* prior adequate trial of Esomeprazole;
* active medical problems such as unstable seizures, or significant physical illness (e.g., serious liver or renal pathology).

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the Social Responsiveness Scale, 2nd Edition (SRS-2) | Baseline, 4 Weeks, 8 Weeks
  Social Responsiveness Scale (SRS) raw scores measure social abilities with lower raw scores meaning better social abilities. (Raw Score Range: 0 - 195)

SECONDARY OUTCOMES:
Change from Baseline on the Aberrant Behavior Checklist, 2nd Edition (ABC-2) | Baseline, 4 Weeks, 8 Weeks
  Higher scores indicate more symptoms, lower scores indicate fewer symptoms. Irritability scores can range from 0-45. Lethargy scores can range from 0-48. Stereotypy scores can range from 0-21. Hyperactivity scores can range from 0-48. Inappropriate speech scores can from 0-12.

OTHER OUTCOMES:
Change from Baseline on the Short Sensory Profile Questionnaire (SSPQ) | Baseline, 4 Weeks, 8 Weeks
Change from Baseline on the Repetitive Behavoiors Scale- Revised (RBS-R) | Baseline, 4 Weeks, 8 Weeks
Change from Baseline on the Stanford Social Motivation Scale (SSMS) | Baseline, 4 Weeks, 8 Weeks
Change from Baseline on the Vineland Adaptive Behavoir Scales - 3 (VABS-3) | Baseline, 4 Weeks, 8 Weeks
Change from Baseline on the Dimensional Assessment of Repetitive Behavior (DARB) | Baseline, 4 Weeks, 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No